CLINICAL TRIAL: NCT06592404
Title: The (Cost)Effectiveness of a Social Robot in Decreasing Professional Caregiver Support and Increasing Independence for Persons in Disability Care Experiencing Problems in Daily Structure and Planning: a Multiple Baseline Case Study
Brief Title: The (Cost)Effectiveness of a Social Robot for Persons with Problems in Daily Structure and Planning in Disability Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academy Het Dorp (Other)
Collaborators: Tilburg University (Other); Maastricht University (Other); KU Leuven (Other); Ipse de Bruggen, disability care organisation (Unknown); SGL, disability care organisation (Unknown); Hartekamp Groep, disability care organisation (Unknown); Disability Studies in Nederland, foundation for disability studies in the Netherlands (Unknown); ZoTeG, academic workplace on technology in disability care (Unknown)
Responsible Party: Principal Investigator, Brigitte Boon, Prof. Dr., Academy Het Dorp
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AHD23.019; 10310012210009 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-07-18; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Brain Injury, Chronic; Intellectual Disability, Mild to Moderate; Autism Spectrum Disorder; Down Syndrome
Keywords: health care technology; disability care; goal attainment; daily structure and planning; social robot; independence
MeSH Terms: conditions — Brain Injury, Chronic; Intellectual Disability; Autism Spectrum Disorder; Down Syndrome

STUDY DESIGN:
Intervention Model Description: This is a multiple baseline single case (MBSC) study, involving individuals receiving long-term disability care and experiencing difficulties in daily structure and planning. Each participant serves as its own control and receives the person-oriented intervention involving a social robot. Participants are randomly assigned to one of four clusters. This randomization determines the duration of three phases during the 13-week study period:
  * Control period (care as usual): 2, 3, 4 or 5 weeks, depending on cluster.
  * Intervention period (start using the robot): 6 weeks.
  * Effect measurement period: 5, 4, 3 or 2 weeks, depending on cluster.
  The study period lasts 13 weeks, with a 2-week follow-up measurement scheduled 6 months after the intervention period. The goal is to integrate the social robot into the participants' care plan, with the intention that they continue using the social robot after the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cluster 1 (Experimental): As explained earlier on, all clusters receive the person-oriented intervention, which involves deploying the social robot on personal goals related to selected activities.
  In this study, randomization determines the duration of study periods.
  For cluster 1, periods are planned as follows:
  * Control: 2 weeks (week 1-2)
  * Intervention: 6 weeks (week 3-8)
  * Effect measurement: 5 weeks (week 9-13)
  * Follow-up: 2 weeks (week 34-35)
  Interventions: Device: Robot Tessa
- Cluster 2 (Experimental): For cluster 2, periods are planned as follows:
  * Control: 3 weeks (week 1-3)
  * Intervention: 6 weeks (week 4-9)
  * Effect measurement: 4 weeks (week 10-13)
  * Follow-up: 2 weeks (week 35-36)
  Interventions: Device: Robot Tessa
- Cluster 3 (Experimental): For cluster 3, periods are planned as follows:
  * Control: 4 weeks (week 1-4)
  * Intervention: 6 weeks (week 5-10)
  * Effect measurement: 3 weeks (week 11-13)
  * Follow-up: 2 weeks (week 36-37)
  Interventions: Device: Robot Tessa
- Cluster 4 (Experimental): For cluster 4, periods are planned as follows:
  * Control: 5 weeks (week 1-5)
  * Intervention: 6 weeks (week 6-11)
  * Effect measurement: 2 weeks (week 12-13)
  * Follow-up: 2 weeks (week 37-38)
  Interventions: Device: Robot Tessa

INTERVENTIONS:
Device: Robot Tessa — Tessa is a small flowerpot shaped robot with two amber LED-lit eyes. The robot is always connected to the power network and internet and speaks reminders at a preset time. These notifications are installed by the user, who can be the professional caregiver or in some cases the participant themselves, using an accessible web app.
  Together with the participant and their professional caregiver, selected activities are translated into goals that the robot will support using Goal Attainment Scaling (Kiresuk & Sherman, 1968), an individualized evaluation method to monitor the progress of (treatment) goals. The goals are evaluated weekly during the study period using a 5-point scale.
  Other Names: Tinybot Tessa

SUMMARY:
The goal of this multiple baseline single case study is to study the (cost)effectiveness of a social robot in reducing professional caregiver support and promoting independence for individuals in long-term disability care experiencing problems with daily structure and planning. The main research questions it aims to answer are:

* What is the effect of the social robot on the frequency of moments professional caregivers support individuals experiencing problems with daily structure and planning with the execution of daily activities, compared to care as usual, after 6 weeks?
* Does the effect of the social robot persist in the long term (after 6 months)?
* What is the cost-effectiveness of the social robot?

Participants will:

* Use a social robot in their daily living environment
* Answer survey questions about their quality of life and wellbeing during the study period
* Share their experiences in interviews

Their profesional caregivers will:

* Register the frequency and duration of support they provide to the participant daily for 13 weeks and a 2-week follow-up
* Give weekly updates and score participants' goal attainment while using the social robot
* Fill in questionnaires on participants' productivity and health care consumption during the study period
* Share their experiences in interviews

DETAILED DESCRIPTION:
Many individuals receiving long-term disability care experience problems in daily structure and planning. This includes people with autism spectrum disorder, mild to moderate intellectual disability, acquired brain injury and/or Down syndrome.

A large number of these individuals need assistance in carrying out daily activities due to these difficulties in planning and organisation. these difficulties include for example being on time for appointments, getting up and going to bed on time, self-care (forgetting to eat or take medication), performing household tasks, and remembering information. Both professional caregivers and clients invest a significant amount of effort, time, and enery into structuring and creating an overview in daily planning.

The use of a social robot that can be programmed to assist with reminders and guidance offers opportunities for both clients and professional caregivers:

* The use of the social robot is expected to lead to more independence and improved well-being for the participant.
* Because the social robot potentially shortens or takes over support moments, professional caregivers might, for example, be deployed more efficiently.
* Positive effects may also be observed in the relationship between professional caregiver and client: when the client functions more independently and their well-being improves, professional caregivers expectedly experience more job satisfaction, which is important for the quality of care and retention of care staff.

The purpose of this study is to research the effectiveness of a social robot in long-term disability care. The study follows participants and their professional caregivers in their daily care setting, first without the social robot (care as usual), then while using the social robot. This study contributes to knowledge about the effective deployment of technology in long-term disability care.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Living in an inpatient long-term disability care facility
* Participant 1) has difficulty with planning and structuring and/or remembering tasks, appointments, and activities, and/or 2) needs outside activation to execute tasks, appointments, and activities
* Able to understand verbal instructions and willing to follow these
* Cognitive capacity to, together with their professional caregiver, set goals to work on with the social robot
* Motivated to work with the social robot on 3-5 goals, for which the participant receives daily or weekly guidance in their home
* Professional caregivers are motivated to participate in the study

Exclusion Criteria:

* Prone to express tension in physical aggression
* Highly sensitive to auditory stimuli

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of professional caregiver support per week | During the whole study period (13 weeks) and 2 weeks follow-up
  This concerns support provided by professional caregivers to the participant regarding the selected activities for which the social robot is used. This support is recorded daily by professional caregivers during the entire study period of 13 weeks and during the two-week follow-up measurement.

SECONDARY OUTCOMES:
Psychosocial impact of technology assessed by PIADS-10 | week 13, follow-up
  Conducted in the form of a structured interview at two moments (effect measurement and follow-up period). The 10-item version of the PIADS (Psychosocial Impact of Assistive Device Scale) measures the impact of the social robot on the ability to adapt to the activities of daily living, ability to participate, ability to take advantage of opportunities, eagerness to try new things, happiness, independence, productivity, quality of life, self-esteem, and sense of control.
Work engagement and added value of the social robot as experienced by professional caregivers | week 13, follow-up
  Based on an interview at two moments (effect measurement and follow-up period) with the professional caregivers. The interview asks about the social robot's effect on work engagement and about the perceived added value of the social robot for each participant from the perspective of the professional caregiver and the added value for the professional caregiver (the pros and cons of using the social robot).
Wellbeing assessed by PWI-ID | Differs per cluster: week 2, week 8, week 9, week 13 (cluster 1); week 3, week 9, week 10, week 13 (cluster 2); week 4, week 10, week 11, week 13 (cluster 3), week 5, week 11, week 12, week 13 (cluster 4), and follow-up (all clusters)
  The PWI-ID (Personal Welbeing Index - Intellectual Disability) is administered five times during the study period. The PWI-ID is designed for people who have an intellectual disability or other form of cognitive impairment. The scale measures eight items, each one corresponding to a quality of life domain: life satisfaction, standard of living, health, life achievement, personal relationships, personal safety, community-connectedness, and future security.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte JF Boon, Prof. Dr., Principal Investigator — Academy Het Dorp, Arnhem, The Netherlands
Locations (3):
- Netherlands (3):
  - SGL, Sittard, Limburg
  - Hartekamp Groep, Velserbroek, North Holland
  - Ipse de Bruggen, Zoetermeer, South Holland